CLINICAL TRIAL: NCT05194475
Title: Metabolic Effects of a Thermogenic Ready-to-drink Beverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: EHP Labs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB2021-676
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Metabolic Rate; Metabolism
Keywords: dietary supplement; energy drink; thermogenic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermogenic Ready-to-drink Beverage (Experimental): Arm in which a thermogenic ready-to-drink beverage is ingested.
  Interventions: Other: Thermogenic Ready-to-drink Beverage
- Placebo Ready-to-drink Beverage (Placebo Comparator): Arm in which a placebo ready-to-drink beverage is ingested.
  Interventions: Other: Placebo Ready-to-drink Beverage

INTERVENTIONS:
Other: Thermogenic Ready-to-drink Beverage — Thermogenic ready-to-drink beverage, which will be ingested by the participant.
  Arms: Thermogenic Ready-to-drink Beverage
Other: Placebo Ready-to-drink Beverage — Placebo ready-to-drink beverage, which will be ingested by the participant.
  Arms: Placebo Ready-to-drink Beverage

SUMMARY:
This study is a randomized, double-blind, placebo-controlled crossover trial examining the metabolic effects of a novel ready-to-drink (RTD) beverage. Healthy adult males and females will be recruited for participation. Each participant will complete two conditions in random order: 1) RTD thermogenic beverage ; and 2) placebo (consisting of the flavoring of the thermogenic beverage without the active ingredients). In each condition, metabolism (resting metabolic rate), hemodynamic (heart rate and blood pressure), and subjective (ratings of energy, focus, concentration, alertness, and mood) assessments will be completed at baseline, 30 minutes after beverage consumption, and 30 minutes after the second round of assessments.

DETAILED DESCRIPTION:
The primary purpose of this study is to report the metabolic effects of a new ready-to-drink (RTD) version of EHP Labs OxyShred Thermogenic Fat Burner. Additionally, the effect of this product on hemodynamic variables and subjective ratings of energy, focus, concentration, alertness, and mood will be reported.

OxyShred Thermogenic Fat Burner (EHP Labs) is a popular dietary supplement for those seeking to increase energy and reduce body fat. While this product is commercially available as a powdered dietary supplement, a new RTD formulation is currently being developed. While the RTD formula will be similar to the current version of the product, research specifically conducted with the RTD version is needed to definitively support product claims and demonstrate the potential effects of this novel product. Additionally, there is a need to better understand the effects of caffeine-containing, thermogenic products among the variety of groups who may consume these products (e.g., males vs. females, inactive vs. active, etc.).

This study is a randomized, double-blind, placebo-controlled crossover trial examining the metabolic effects of a novel ready-to-drink (RTD) beverage. Healthy adult males and females will be recruited for participation. Each participant will complete two conditions in random order: 1) RTD thermogenic beverage ; and 2) placebo (consisting of the flavoring of the thermogenic beverage without the active ingredients). In each condition, metabolism (resting metabolic rate), hemodynamic (heart rate and blood pressure), and subjective (ratings of energy, focus, concentration, alertness, and mood) assessments will be completed at baseline, 30 minutes after beverage consumption, and 30 minutes after the second round of assessments.

ELIGIBILITY:
The inclusion criteria are:

* Between the ages of 18 and 40.
* Body mass between 50 - 110 kg (110 - 220 lbs.).
* Either: (A) Resistance-trained, defined as completing 3+ resistance training sessions per week for at least two years prior to screening; full body (all upper body and lower body major muscle groups) must be trained at least once weekly, OR (B) non-resistance trained, defined as never having followed a structured resistance training program.
* Perform ≤ 30 minutes of high-intensity interval training per week.
* Perform ≤ 60 minutes of steady state endurance exercise per week.
* Regular caffeine consumption (due to the presence of caffeine in the commercially available dietary supplement). This will be defined as an average self-reported daily intake of 200+ mg of caffeine, which is equivalent to approximately 2 cups of coffee.

The exclusion criteria are:

* Failing to meet any of the aforementioned inclusion criteria.
* Presence of any known disease or medical condition which could be negatively affected by consumption of the beverage. This includes cardiovascular disease or condition; liver disease or disorder; other metabolic disease or disorder; or other conditions that could reasonably be deemed to contraindicate the study protocol.
* Pregnant or breastfeeding, based on self-report (for female participants).
* Taking medication which could reasonably make participation unsafe for the participant or influence study outcomes. Specifically, use of any prescription stimulant (e.g., dextroamphetamine (Dexedrine®), dextroamphetamine/amphetamine combination product (Adderall®), methylphenidate (Ritalin®, Concerta®), or similar stimulants) precludes participation in this study.
* Self-reported caffeine sensitivity, as indicated by unwanted side effects when caffeine is consumed.
* Allergy to any of the ingredients in the RTD beverage.
* Presence of a pacemaker or other implanted electrical device
* Self-reported claustrophobia (due to metabolism testing)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Resting metabolic rate | 140 minutes
  Resting metabolic rate from indirect calorimetry expressed as kilocalories expended per unit time (e.g., kcal/min).
Respiratory quotient | 140 minutes
  Respiratory quotient from indirect calorimetry in arbitrary units, which reflects the proportion of carbohydrate and fat oxidized at rest.

SECONDARY OUTCOMES:
Subjective rating of energy | 140 minutes
  Subjective rating of energy as assessed by visual analog scale.
Subjective rating of focus | 140 minutes
  Subjective rating of focus as assessed by visual analog scale.
Subjective rating of concentration | 140 minutes
  Subjective rating of concentration as assessed by visual analog scale.
Subjective rating of alertness | 140 minutes
  Subjective rating of alertness as assessed by visual analog scale.
Subjective rating of mood | 140 minutes
  Subjective rating of mood as assessed by visual analog scale.
Heart rate | 140 minutes
  Heart rate from automated sphygmomanometer expressed in beats per minute.
Systolic blood pressure | 140 minutes
  Systolic blood pressure from automated sphygmomanometer expressed in beats per minute.
Diastolic blood pressure | 140 minutes
  Diastolic blood pressure from automated sphygmomanometer expressed in beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Grant M Tinsley, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Department of Kinesiology & Sport Management, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided